CLINICAL TRIAL: NCT04808765
Title: Experience and Comparison Between Closed Incision Disposable Negative Pressure Wound Therapy With Standard Care in Immediate Postmastectomy Breast Reconstruction - Prospective, Randomized and Controlled Study
Brief Title: Closed Incision Disposable Negative Pressure Wound Therapy in Immediate Postmastectomy Breast Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University in Zielona Góra (Other)
Collaborators: ConvaTec Inc. (Industry)
Responsible Party: Principal Investigator, Karolina Pieszko, Principal Investigator, University in Zielona Góra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZG01012019
Record Dates: First submitted 2021-03-17; First posted 2021-03-22 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer; Breast Reconstruction
Keywords: breast cancer; closed incision negative pressure wound therapy; Breast Reconstruction
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammaplasty; Drug Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VAC group (Experimental): A randomized group of patients receiving negative pressure wound therapy dressing (Avelle-ConvaTec) on closed incision
  Interventions: Procedure: Immediate Breast reconstruction
- ST group (Active Comparator): A randomized group of patients receiving standard dressing (sterile gauze and medical tape) on closed incision
  Interventions: Procedure: Immediate Breast reconstruction

INTERVENTIONS:
Procedure: Immediate Breast reconstruction — immediate mastectomy with breast reconstruction with implants or expanders
  Other Names: immediate mastectomy with breast reconstruction with implants or expanders

SUMMARY:
The study aimed to assess the impact of the use of closed incision negative pressure wound therapy (ciNPWT) after immediate breast reconstruction on the number of surgical-site complications, skin surface temperature, objective elastic and viscoelastic and subjective scar's quality to determine risk factors that could be considered as indications for prophylactic ciNPWT application.

DETAILED DESCRIPTION:
Breast cancer excluding skin cancer is the most commonly diagnosed cancer after lung cancer among women. In recent years, the incidence rate of breast cancer has been rising by 0,3% annually. Screening tests are designed to diagnose breast cancer in possible early stadium of disease. Rapid diagnosis and efficacy of neoadjuvant and adjuvant therapies influence on immediate breast reconstructions after skin (SSM) and nipple-sparing mastectomies (NSM). The prophylactic methods of reducing a higher wound healing complication rate after neoadjuvant and adjuvant therapies are crucial.

The study aimed to assess the impact of the use of closed incision negative pressure wound therapy (ciNPWT) after immediate breast reconstruction on the number of surgical-site complications, skin surface temperature, objective elastic and viscoelastic and subjective scar's quality to determine risk factors that could be considered as indications for prophylactic ciNPWT application.

The analysis included data from anamnesis, details of performed surgical procedure, measurements of skin surface temperature with Skin-Thermometer® probe, measurements of skin elasticity with Cutometer® probe, and scar assessments according to POSAS v2.0 questionnaire for patient and observer.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years of age
* indications for immediate breast reconstruction

Exclusion Criteria:

* pregnancy or lactation,
* use of steroids, use of immune modulators known to affect wound healing;
* tattoos in the area of the incision;
* breast skin conditions such as cutis laxa;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female patients with indications for immediate breast reconstruction
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Postsurgical complications - reported for 60 patients | 1 month
  surgical site complications
Postsurgical complications - reported for 60 patients | 1 year
  surgical site complications

SECONDARY OUTCOMES:
Superficial Skin Temperature (SST) of scar, skin next to scar and the second breast | 1 week after surgery
  measure SST with Skin-Thermometer
Superficial Skin Temperature (SST) of scar, skin next to scar and the second breast | 1 month after surgery
  measure SST with Skin-Thermometer
Objective examination of scar quality | 1 year after surgery
  measure skin elasticity with Cutometer
Subjective examination of scar quality | 1 year after surgery
  POSAS 2.0 (Patient and Observer Scar Assessment Scale) questionnaire for the observer and the patient.
  Questions regards painful, itchy scar, difference between scar and normal skin. The min score is 7, the max score is 70. The higher score means better result
Subjective quality of life | 1-2 years after surgery
  BREAST-Q reconstruction module and Breast implant illness survey for patients. Questions about self-confidence, comfort, acceptance of new appearance, feeling of implants, breast pain. The min score is 1, the max 3-5 depending on part of questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Dawid Murawa, PROF, Study Chair — University in Zielona Gora
Locations (1):
- University in Zielona Gora, Zielona Góra, Lubusz Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Singh D, Lobach V, Holton T. Use of Closed-Incision Negative-Pressure Therapy in Aesthetic Surgery. Plast Reconstr Surg. 2019 Jan;143(1S Management of Surgical Incisions Utilizing Closed-Incision Negative-Pressure Therapy):11S-14S. doi: 10.1097/PRS.0000000000005306. PMID 30586097
- [Result] Willy C, Agarwal A, Andersen CA, Santis G, Gabriel A, Grauhan O, Guerra OM, Lipsky BA, Malas MB, Mathiesen LL, Singh DP, Reddy VS. Closed incision negative pressure therapy: international multidisciplinary consensus recommendations. Int Wound J. 2017 Apr;14(2):385-398. doi: 10.1111/iwj.12612. Epub 2016 May 12. PMID 27170231
- [Result] Gabriel A, Sigalove SR, Maxwell GP. Initial Experience Using Closed Incision Negative Pressure Therapy after Immediate Postmastectomy Breast Reconstruction. Plast Reconstr Surg Glob Open. 2016 Jul 22;4(7):e819. doi: 10.1097/GOX.0000000000000803. eCollection 2016 Jul. PMID 27536498
- [Result] Gabriel A, Sigalove S, Sigalove N, Storm-Dickerson T, Rice J, Maxwell P, Griffin L. The Impact of Closed Incision Negative Pressure Therapy on Postoperative Breast Reconstruction Outcomes. Plast Reconstr Surg Glob Open. 2018 Aug 7;6(8):e1880. doi: 10.1097/GOX.0000000000001880. eCollection 2018 Aug. PMID 30324063